CLINICAL TRIAL: NCT00990600
Title: Adherence to a One Pill, Once-a-day Antiretroviral Regimen
Brief Title: QoL and Adherence to One-pill Once-a-day HAART
Acronym: ADONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Franco Maggiolo MD, Divisione di Malattie Infettive, Ospedali Riuniti, Bergamo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADONE; EUDRACT NUMBER: 2007-007839-33
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: HIV Infection; HIV Infections
Keywords: adherence; Qol; virologic efficacy; immunologic efficacy; patients' preference; once-daily; HAART; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simplified one pill regimen (Experimental): Fixed dose combination of tenofovir + emtricitabine + efavirenz
  Interventions: Other: reduced number of pills

INTERVENTIONS:
Other: reduced number of pills — Switch to a fixed dose combination one pill/daily HAART
  Other Names: efavirenz EFV; emtricitabine FTC; tenofovir TDF

SUMMARY:
Primary objective of the study is:

To verify if simplification of the antiretroviral regimen, measured as the reduction of pill burden alone, may affect adherence rate of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent signed
* Effective ongoing treatment (HIV-RNA < 50 copies/ml) for at least three months
* Being on a stable HAART regimen based either on two possible drug associations:

  * 3TC/FTC + TDF + EFV
  * FTC/TDF (fixed dose combination) + EFV
* No previous documented virologic failure

Exclusion Criteria:

* Childbearing or breastfeeding. Women of childbearing potential will be asked to adopt effective contraceptive methods or behaviours
* Any ongoing grade 4 laboratory abnormality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Proportion of adherence to HAART | 6 months

SECONDARY OUTCOMES:
QoL (VAS scale) preferences of patients virologic and immunologic outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Maggiolo, MD, Principal Investigator — Ospedali Riuniti, Bergamo